CLINICAL TRIAL: NCT04151017
Title: Efficacy of Autologous Fibrin Glue Versus Suture for Conjuntival Autografting in Primary Pterygium Surgery: a Randomized Clinical Trials
Brief Title: Efficacy of Autologous Fibrin Glue in Pterygium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170467
Record Dates: First submitted 2019-09-27; First posted 2019-11-05 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous fibrin glue (Experimental)
  Interventions: Other: Autologous fibrin glue
- Sutures (Active Comparator)
  Interventions: Other: Suture

INTERVENTIONS:
Other: Autologous fibrin glue — Conjunctival graft fixation with autologous fibrin glue
  Arms: Autologous fibrin glue
Other: Suture — Graft fixation using 10.0 mononylon
  Arms: Sutures

SUMMARY:
Pterygium is wing-shaped, vascular, fleshy growth that originates on the conjuntiva and that can spread to the corneal limbus and beyond The surgical exeresis with autologous conjunctival autograft technique is the treatment of choice. Commercially available fibrin glue has been used preferentially for graft fixation due to its benefits compared to sutures; However, its cost and the risk of inflammatory immune reaction limit the its use. There are few studies about autologous fibrin glue.

OBJECTIVE: To determine the efficacy of autologous fibrin glue preparation in patients undergoing pterygium resection surgery. To compare with autologous conjunctival graft fixation with suture.

This is a randomized clinical trial. Two patient groups will undergo pterygium excision surgery. Group 1 will have autologous conjunctival graft fixation with autologous fibrin glue and group 2 will have suture graft fixation using 10.0 mononylon. Early and late postoperative surgical results as well as complication rates will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* nasal primary pterygium

Exclusion Criteria:

* relapsed pterygium
* patients with a history of previous eye surgery
* patients with glaucoma using hypotensive eye drops
* eye surface diseases
* eye allergy
* diabetic patients,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pterygium Recurrence | 6 months
  Recurrence in 6 months

SECONDARY OUTCOMES:
Autograft Retraction | Postoperative day 1, 7, 21 and 30
  Graft detachment or retraction
Postoperative Pain | Postoperative day 1, 7, 21 and 30
  Presence Pain measured by a five-point scale, in which 0 means absence of symptom; 1 means easily tolerable symptom; 2 means symptom causing some discomfort; 3 means symptom partially interfering with usual activities and 4 means symptom completely interfering with usual activities
Graft Edema | Postoperative day 1, 7, 21 and 30
  Graft edema (1-4).

CONTACTS AND LOCATIONS:
Overall Officials: Diane Marinho, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Santa Casa de Misericórdia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cioba C, Marafon SB, Fortes BGB, Cavalheiro MT, Fabris M, Michel G, Zambon GM, Marcon A, Marinho DR. Autologous fibrin glue versus sutures for conjunctival autograft in primary pterygium: a randomized clinical trial. Int Ophthalmol. 2023 Jul;43(7):2371-2381. doi: 10.1007/s10792-023-02635-z. Epub 2023 Jan 18. PMID 36652022